CLINICAL TRIAL: NCT05390294
Title: Prognostic Factors for Survival of Patients With Salivary Gland Malignancies
Brief Title: Survival With Patients Treated With Salivary Gland Cancer
Status: Completed | Type: Observational
Sponsor: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, Denis Brajković, Principal Investigator, Clinical Center of Vojvodina
Other Study IDs: 1106012
Record Dates: First submitted 2022-05-18; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Salivary Gland Cancer; Salivary Gland Neoplasms
Keywords: Salivary gland cancer; Survival; Prognostic factors
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients free of the disease: Patients treated due to SGC without local recurrence or metastases
  Interventions: Procedure: Surgical intervention with or without postoperative adjuvant therapy
- Patients with the disease: Patient with relapse of SGC, metastases or died due to SGC
  Interventions: Procedure: Surgical intervention with or without postoperative adjuvant therapy

INTERVENTIONS:
Procedure: Surgical intervention with or without postoperative adjuvant therapy — Surgical intervention with or without postoperative adjuvant therapy

SUMMARY:
Salivary gland malignancies is very heterogenous group of tumors regarding tumor histology and localization. The aim of this study is to assess main clinical and pathological parameters related to patients survival

DETAILED DESCRIPTION:
The retrospective study enrolled medical charts of the patients treated due to salivaly gland cancers in the Clinic for maxillofacial surgery at Clinical center of Vojvodina in the period of 1. January 1996. to 31. December 2021. Patients demographics, type of the tumor, localization, TNM status and patohystological parameters were evaluated for patients survival and disease free periods

ELIGIBILITY:
Inclusion Criteria:

Patients with salivary gland malignancies treted in the Clinic for maxillofacial surgery

Exclusion Criteria:

Incomplete medical data Patients with metastatic tumord of salivary gland Patients with recurrent malignancies of salivary glands sent from other clinics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated due to SGC in the Clinic for maxillofacial surgery at Clinical center of Vojvodina
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Patients survival | Through study completion, an average of 1 year
  Survival of patients treated due to SGC during observation period of minimum 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for maxillofacial surgery Clinical center of Vojvodina, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: No